CLINICAL TRIAL: NCT06337552
Title: A Randomized High-Fermented Food Intervention Among Locally Advanced Rectal Cancer Patients (The FEED Trial)
Brief Title: High-Fermented Food Intervention Among Locally Advanced Rectal Cancer Patients (The FEED Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCC-22709
Record Dates: First submitted 2024-03-18; First posted 2024-03-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Rectal Cancer; Non-Small Cell Lung Cancer
Keywords: Locally Advanced; Rectal Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Rectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the FEED-FF Arm or the Standard of Care (SUC) Arm
Who Masked: Care Provider
Masking Description: Clinical response will be determined in clinic when patients undergo blinded tumor assessments by standard digital rectal exam, endoscopy, and rectal MRI at baseline and at the end of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FEED-FF (Experimental): Participants will be asked to pick up the fermented foods at the Research Kitchen at Moffitt. Participants will be asked to eat 3-6 servings of FFs per day, from 1 week prior to treatment start through 12 weeks after treatment start/until the restaging scope is completed.
  At baseline, the end of week 6.5 and again at week 12.5, participants will be asked to provide biospecimens including a stool sample collected at home and a blood specimen collected in clinic.
  Participants will be asked to complete a food frequency questionnaire, a quality-of-life survey, two symptom related surveys, and a stool collection questionnaire at these same timepoints.
  After the dietary intervention, participants will be asked to complete an exit survey to provide feedback on the study and intervention.
  Interventions: Other: FEED-FF
- Standard of Care (SUC) (Active Comparator): Participants will receive general healthy eating handouts similar to current usual care documents provided in clinic.
  These handouts will detail typical healthy foods and the suggested level of intake, or servings per day.
  At baseline, the end of week 6.5 and again at week 12.5, participants will be asked to provide biospecimens including a stool sample collected at home and a blood specimen collected in clinic. Participants will be asked to complete a food frequency questionnaire, a quality-of-life survey, two symptom related surveys, and a stool collection questionnaire at these same timepoints.
  Interventions: Other: Standard of Care (SUC)

INTERVENTIONS:
Other: FEED-FF — 3-6 servings of any combination of the following fermented foods/day (from 1 week prior to treatment to approximately 12 weeks after the start of treatment): Yogurt, cottage cheese, kefir, kombucha, sauerkraut, and kimchi.
  Arms: FEED-FF
Other: Standard of Care (SUC) — Standard of Care (SUC) is the treatment that is accepted by medical experts as a proper treatment for a certain type of disease and that is widely used by health care professionals. Standard of Care will comprise general healthy eating handouts that describe typical healthy foods and the suggested level of servings per day.
  Arms: Standard of Care (SUC)

SUMMARY:
The purpose of the study is to evaluate the feasibility and acceptability of a dietary intervention (FEED-FF) that includes fermented foods (FF), among locally advanced rectal cancer patients and non-small cell lung cancer (NSCLC) patients, and to explore whether this diet can improve outcomes in rectal cancer patients receiving chemoradiation and NSCLC patients receiving immunotherapy.

ELIGIBILITY:
Inclusion Criteria for GI Patients:

* 18 years of age or older
* Diagnosed with locally advanced rectal cancer (Stage II-III)
* Will undergo neoadjuvant chemoradiation at Moffitt Cancer Center
* Able to pick up FFs once/weekly at Moffitt
* Able to speak and read English
* Able to consume foods orally
* Able to provide informed consent

Inclusion Criteria for Thoracic Patients:

* 18 years of age or older
* Diagnosed with stage II-IV non-small cell lung cancer (NSCLC)
* Will undergo Immunotherapy with immune checkpoint inhibitors (+/- chemotherapy or other treatment) at Moffitt Cancer Center
* Able to pick up FFs once/weekly at Moffitt
* Able to speak and read English
* Able to consume foods orally
* Able to provide informed consent

Exclusion Criteria:

* Antibiotic use within 1 month prior to baseline
* If currently using probiotics, unwillingness to cease probiotic use
* Previous receipt of surgery, immunotherapy, chemotherapy, or radiation for a colon or rectal tumor
* Per clinician's discretion, clinician confirmed inflammatory bowel conditions (e.g., ulcerative colitis, Crohn's disease)
* Infectious disease diagnosed <1 month prior to baseline
* Already consuming ≥2 servings of fermented foods/day
* Previously diagnosed with a mast cell disorder or histamine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Effects of the FEED-FF diet on clinical response to chemoradiation (Rectal Cancer Patients) | At Baseline and Up to 12.5 Weeks
  Clinical response measured in clinic by MRI/Endoscopy/Digital rectal exam, comparing the FEED-FF arm to SUC arm.
  Indicators of clinical response are Complete Response, Near Complete Response, Incomplete Response, or Progressive Disease.
Effects of the FEED-FF diet on clinical response to immunotherapy (Lung Cancer Patients) | At Baseline and Up to 12.5 Weeks
  Clinical benefit to immune checkpoint inhibitor therapy will be measured in clinic by MRI/Endoscopy, comparing the FEED-FF arm to SUC arm.
  Defined as the best response of complete tumor resolution (CR), Partial Response (PR), and stable tumor size (SD) within 12 months.
  Progressive Disease (PD) within 12 months indicates no clinical benefit.
Effects of FEED-FF diet on the gut microbiome | At Baseline, Week 6.5 and Up to 12.5 Weeks
  Measured by fecal biospecimen sample collection; FEED-FF arm hypothesized to demonstrate increases in short chain fatty acid (SCFA) producing bacteria and higher alpha diversity compared to SUC arm.
Effects of FEED-FF diet on local immune-related biomarkers | At Baseline and Up to 12.5 Weeks
  Measured by FFPE tissue slides; FEED-FF arm hypothesized to demonstrate enhanced immune response such as higher T-cell expression compared to SUC arm.
Effects of FEED-FF diet on quality of life | At Baseline, Week 6.5 and Up to 12.5 Weeks
  Measured by using the European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life (QoL) Survey; FEED-FF arm hypothesized to demonstrate more favorable QoL compared to SUC arm.
Efficacy of the FEED-FF intervention | At Baseline, Week 6.5 and Up to 12.5 Weeks
  Measured by an accrual rate of 50% of eligible patients, fermented foods (FF) intake of at least 3 servings on at least 80% of days, and at least 80% of intervention group reporting high/very high satisfaction with intervention.
  Weekly goal adherence via randomly administered food logs, tracking responses to and general completion of an exit survey will be utilized.
Feasibility of the FEED-FF intervention | At Baseline, Week 6.5 and Up to 12.5 Weeks
  Measured by an accrual rate of 50% of eligible patients, fermented foods (FF) intake of at least 3 servings on at least 80% of days, and at least 80% of intervention group reporting high/very high satisfaction with intervention.
  Weekly goal adherence via randomly administered food logs, tracking responses to and general completion of an exit survey will be utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Doratha (Armen) Byrd, PhD, MPH, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org/clinical-trials-research/clinical-trials/